CLINICAL TRIAL: NCT02018549
Title: An Open Label Placebo Study To Assess The Inhalation Profile Obtained By Acoustic Monitoring In COPD Patients Using The NEXThaler Dry Powder Inhaler (DPI) Device
Brief Title: An Open Label Placebo Study To Assess The Inhalation Profile Obtained By Acoustic Monitoring In COPD Patients Using The NEXThaler DPI
Acronym: PIF3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCD_01535BC1_01; 2013-000262-11 (EudraCT Number)
Record Dates: First submitted 2013-07-03; First posted 2013-12-23 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: COPD
Keywords: COPD; placebo; inhalatory profile
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo (Experimental): Inhalation through Chiesi NEXThaler DPI containing Placebo Dry Powder. Each patient will perform at least two inhalations using the Chiesi NEXThaler DPI device containing placebo dry powder. There is no comparator and all patients will receive the same study treatment.
  Interventions: Device: Inhalation through Chiesi NEXThaler DPI

INTERVENTIONS:
Device: Inhalation through Chiesi NEXThaler DPI — Inhalatory manoeuvre through Chiesi NEXThaler DPI repeated at least twice in order to have two evaluable data set

SUMMARY:
Phase IIa, single center, open-label, single-arm study, to evaluate the inspiration profile through the NEXThaler device in adult COPD patients with varying degrees of airflow limitation

DETAILED DESCRIPTION:
As this is an exploratory study, a total of 70 to 80 completed patients, ensuring the following distribution in terms of COPD Stage as per GOLD 2013 (updated) spirometric classification of disease severity, are deemed to be sufficient for assessing the inhalation profile through the NEXThaler®:

* 10 to 20 COPD GOLD Stage I patients
* 20 patients in each of the COPD GOLD Stage II to IV. Assuming a screening failure/drop-out rate of 10%, a maximum of 89 patients will be screened in order to reach the required number of completed patients.

All the analyses will be performed separately for the first and the second inhalation. Results stratified by disease severity and overall will be presented.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient and/or the legal representatives
2. Inpatients and outpatients of both sexes, aged ≥ 40 years
3. Documented clinical diagnosis (within the past 6 months) of COPD with varying degrees of airflow limitation based on Spirometric classification of disease severity according to GOLD 2013 (updated) guidelines with a smoking history of at least 10 pack years (pack-years = the number of cigarette packs per day times the number of years). Current smokers and ex-smokers are eligible
4. A cooperative attitude and ability to use DPIs and to be trained in the proper use of the NEXThaler® as confirmed by the activation of the training device BAM

Exclusion Criteria:

1. Pregnant women confirmed by a positive pregnancy test or nursing (lactating) women (if applicable)
2. Diagnosis of asthma
3. Diagnosis of restrictive lung disease
4. Allergy to any component of the placebo treatment
5. Inability to comply with study procedures or treatment
6. Significant unstable medical history of and/or treatments for cardiac, renal, neurological, hepatic, endocrine diseases, or any previously documented laboratory abnormality indicative of a significant underlying condition, that may interfere with patient's safety, compliance, or study evaluations, according to the investigator's opinion.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of Inhalatory Profile for 80 patients | Visit 1
  The study duration per patient is only one visit. At visit 1 the patient after having signed the ICF and after having assessed the eligibility criteria should perform two evaluable inhalatory manoeuvres through the device instrumented with an acoustic monitoring system (microphone). The sounds captured by the microphone are sent to a PC which acquire it for analysis of the profile. Each manoeuvre lasts few seconds. After having completed the manoeuvres and have the same assessed as good by the Investigator, the study is completed. All the procedures are expected to be performed within a couple of hours for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Scuri, MD, Study Director — Chiesi Farmaceutici S.p.A.
Locations (1):
- Ospedale di Parma, Parma, Italy

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2013-000262-11
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/CSR_Synopsis_CCD-01535BC1-01.pdf